CLINICAL TRIAL: NCT01567787
Title: Spinal Tumor Proton Protocol
Brief Title: Proton Radiation Therapy for Spinal Tumors
Acronym: NF01
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 1101-NF01
Record Dates: First submitted 2012-03-13; First posted 2012-03-30 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Nerve Sheath Tumors; Neurofibroma
Keywords: Proton Radiation Therapy; Spinal tumors; Neurofibroma(NF1); Malignant peripheral nerve sheath tumor(MPNST)
MeSH Terms: conditions — Nerve Sheath Neoplasms; Neurofibroma; Spinal Cord Neoplasms; Neurofibrosarcoma | interventions — Neurofibromin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proton Radiation for MPNST (Experimental): Proton radiation 30 cobalt gray equivalent(CGE)at 6 CGE per fraction
  Interventions: Radiation: Proton Radiation for MPNST
- Proton Radiation for neurofibromas (Experimental): Proton radiation 25 cobalt gray equivalent(CGE) at 5 CGE per fraction
  Interventions: Radiation: Proton Radiation for neurofibromas

INTERVENTIONS:
Radiation: Proton Radiation for MPNST — 30 CGE at 6 CGE/Fx
  Arms: Proton Radiation for MPNST
Radiation: Proton Radiation for neurofibromas — 25 CGE at 5 CGE/Fx
  Arms: Proton Radiation for neurofibromas

SUMMARY:
The purpose of this study is to determine if Proton Therapy can provide effective and safe treatment for Malignant Peripheral Nerve Sheath Tumors of the spine and Neurofibromas of the spine.

DETAILED DESCRIPTION:
Proton therapy may provide the benefits of local control or palliation, while reducing the risk associated with photon radiation, by delivering therapeutic doses to a well-defined target area with significant reduction in the integral dose. A dosimetry comparison of protons and photons at the University of Florida Proton Therapy Institute confirmed the feasibility of proton irradiation of these tumors with less exposure of normal tissue to radiation than expected with photon techniques. This reduced radiation exposure to uninvolved normal tissues is expected to decrease the risk of radiation-induced second malignancies and neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* MPNSTs that are biopsy-positive and resected, subtotally resected or unresectable.
* Symptomatic (pain, numbness, or weakness) NF1 neurofibromas that are biopsy-positive and unresectable or subtotally resected.
* Symptomatic NF1 neurofibromas that are unbiopsied and PET-negative, if the patient refuses biopsy/surgery or is medically inoperable.
* Asymptomatic NF1 neurofibromas with radiologic progression after surgery.
* PET-positive, unbiopsied lesions in NF1 patients who refuse biopsy/surgery or are medically inoperable.

Exclusion Criteria:

* Spinal instability.
* Metal stabilization hardware within the target area.
* Previously irradiated at this disease site.
* Spinal cord compression with complete loss of function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Local Control | 7 years after completion of RT

SECONDARY OUTCOMES:
Progression or palliation of pain, numbness, or weakness | At 3, 6, 12, 24 and 60 months after RT
Number of adverse events | At 3, 6, 12, 24, 60 months and 15 years after RT
Quality of Life | 3, 6, 12, 24 and 60 months after RT
Rate of malignant transformation within the high-dose volume | 15 years after RT
Rate of second malignant primaries outside of high dose volume, but located in tissues exposed to radiation within the beam path | 15 years after RT

CONTACTS AND LOCATIONS:
Overall Officials: Randal H Henderson, MD, Principal Investigator — University of Florida Proton Therapy Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hottinger AF, Khakoo Y. Neuro-oncology of Neurofibromatosis Type 1. Curr Treat Options Neurol. 2009 Jul;11(4):306-14. doi: 10.1007/s11940-009-0034-4. PMID 19523356
- [Background] Friedman JM, Birch PH. Type 1 neurofibromatosis: a descriptive analysis of the disorder in 1,728 patients. Am J Med Genet. 1997 May 16;70(2):138-43. doi: 10.1002/(sici)1096-8628(19970516)70:23.0.co;2-u. PMID 9128932
- [Background] Cnossen MH, de Goede-Bolder A, van den Broek KM, Waasdorp CM, Oranje AP, Stroink H, Simonsz HJ, van den Ouweland AM, Halley DJ, Niermeijer MF. A prospective 10 year follow up study of patients with neurofibromatosis type 1. Arch Dis Child. 1998 May;78(5):408-12. doi: 10.1136/adc.78.5.408. PMID 9659085
- [Background] Mautner VF, Asuagbor FA, Dombi E, Funsterer C, Kluwe L, Wenzel R, Widemann BC, Friedman JM. Assessment of benign tumor burden by whole-body MRI in patients with neurofibromatosis 1. Neuro Oncol. 2008 Aug;10(4):593-8. doi: 10.1215/15228517-2008-011. Epub 2008 Jun 17. PMID 18559970
- [Background] Seppala MT, Haltia MJ, Sankila RJ, Jaaskelainen JE, Heiskanen O. Long-term outcome after removal of spinal neurofibroma. J Neurosurg. 1995 Apr;82(4):572-7. doi: 10.3171/jns.1995.82.4.0572. PMID 7897516
- [Background] Thakkar SD, Feigen U, Mautner VF. Spinal tumours in neurofibromatosis type 1: an MRI study of frequency, multiplicity and variety. Neuroradiology. 1999 Sep;41(9):625-9. doi: 10.1007/s002340050814. PMID 10525761
- [Background] Tonsgard JH. Clinical manifestations and management of neurofibromatosis type 1. Semin Pediatr Neurol. 2006 Mar;13(1):2-7. doi: 10.1016/j.spen.2006.01.005. PMID 16818170
- [Background] Needle MN, Cnaan A, Dattilo J, Chatten J, Phillips PC, Shochat S, Sutton LN, Vaughan SN, Zackai EH, Zhao H, Molloy PT. Prognostic signs in the surgical management of plexiform neurofibroma: the Children's Hospital of Philadelphia experience, 1974-1994. J Pediatr. 1997 Nov;131(5):678-82. doi: 10.1016/s0022-3476(97)70092-1. PMID 9403645
- [Background] Ducatman BS, Scheithauer BW, Piepgras DG, Reiman HM, Ilstrup DM. Malignant peripheral nerve sheath tumors. A clinicopathologic study of 120 cases. Cancer. 1986 May 15;57(10):2006-21. doi: 10.1002/1097-0142(19860515)57:103.0.co;2-6. PMID 3082508
- [Background] Evans DG, Baser ME, McGaughran J, Sharif S, Howard E, Moran A. Malignant peripheral nerve sheath tumours in neurofibromatosis 1. J Med Genet. 2002 May;39(5):311-4. doi: 10.1136/jmg.39.5.311. PMID 12011145
- [Background] Ferner RE, Gutmann DH. International consensus statement on malignant peripheral nerve sheath tumors in neurofibromatosis. Cancer Res. 2002 Mar 1;62(5):1573-7. PMID 11894862
- [Background] Chao RC, Pyzel U, Fridlyand J, Kuo YM, Teel L, Haaga J, Borowsky A, Horvai A, Kogan SC, Bonifas J, Huey B, Jacks TE, Albertson DG, Shannon KM. Therapy-induced malignant neoplasms in Nf1 mutant mice. Cancer Cell. 2005 Oct;8(4):337-48. doi: 10.1016/j.ccr.2005.08.011. PMID 16226708
- [Background] Stiller CA, Chessells JM, Fitchett M. Neurofibromatosis and childhood leukaemia/lymphoma: a population-based UKCCSG study. Br J Cancer. 1994 Nov;70(5):969-72. doi: 10.1038/bjc.1994.431. PMID 7947106
- [Background] Huson SM, Compston DA, Harper PS. A genetic study of von Recklinghausen neurofibromatosis in south east Wales. II. Guidelines for genetic counselling. J Med Genet. 1989 Nov;26(11):712-21. doi: 10.1136/jmg.26.11.712. PMID 2511319
- [Background] Sharif S, Ferner R, Birch JM, Gillespie JE, Gattamaneni HR, Baser ME, Evans DG. Second primary tumors in neurofibromatosis 1 patients treated for optic glioma: substantial risks after radiotherapy. J Clin Oncol. 2006 Jun 1;24(16):2570-5. doi: 10.1200/JCO.2005.03.8349. PMID 16735710
- [Background] Papageorgio C, Seiter K, Feldman EJ. Therapy-related myelodysplastic syndrome in adults with neurofibromatosis. Leuk Lymphoma. 1999 Feb;32(5-6):605-8. doi: 10.3109/10428199909058420. PMID 10048435
- [Background] Gerszten PC, Burton SA, Ozhasoglu C, McCue KJ, Quinn AE. Radiosurgery for benign intradural spinal tumors. Neurosurgery. 2008 Apr;62(4):887-95; discussion 895-6. doi: 10.1227/01.neu.0000318174.28461.fc. PMID 18496194
- [Background] Karabatsou K, Kiehl TR, Wilson DM, Hendler A, Guha A. Potential role of 18fluorodeoxyglucose-positron emission tomography/computed tomography in differentiating benign neurofibroma from malignant peripheral nerve sheath tumor associated with neurofibromatosis 1. Neurosurgery. 2009 Oct;65(4 Suppl):A160-70. doi: 10.1227/01.NEU.0000337597.18599.D3. PMID 19927062
- [Background] Ferner RE, Golding JF, Smith M, Calonje E, Jan W, Sanjayanathan V, O'Doherty M. [18F]2-fluoro-2-deoxy-D-glucose positron emission tomography (FDG PET) as a diagnostic tool for neurofibromatosis 1 (NF1) associated malignant peripheral nerve sheath tumours (MPNSTs): a long-term clinical study. Ann Oncol. 2008 Feb;19(2):390-4. doi: 10.1093/annonc/mdm450. Epub 2007 Oct 11. PMID 17932395
- [Background] Warbey VS, Ferner RE, Dunn JT, Calonje E, O'Doherty MJ. [18F]FDG PET/CT in the diagnosis of malignant peripheral nerve sheath tumours in neurofibromatosis type-1. Eur J Nucl Med Mol Imaging. 2009 May;36(5):751-7. doi: 10.1007/s00259-008-1038-0. Epub 2009 Jan 14. PMID 19142634
- [Background] Wentworth S, Pinn M, Bourland JD, Deguzman AF, Ekstrand K, Ellis TL, Glazier SS, McMullen KP, Munley M, Stieber VW, Tatter SB, Shaw EG. Clinical experience with radiation therapy in the management of neurofibromatosis-associated central nervous system tumors. Int J Radiat Oncol Biol Phys. 2009 Jan 1;73(1):208-13. doi: 10.1016/j.ijrobp.2008.03.073. Epub 2008 Aug 5. PMID 18687535
- [Background] Chopra R, Morris CG, Friedman WA, Mendenhall WM. Radiotherapy and radiosurgery for benign neurofibromas. Am J Clin Oncol. 2005 Jun;28(3):317-20. doi: 10.1097/01.coc.0000156923.52181.3d. PMID 15923807
- [Background] Sahgal A, Chou D, Ames C, Ma L, Lamborn K, Huang K, Chuang C, Aiken A, Petti P, Weinstein P, Larson D. Image-guided robotic stereotactic body radiotherapy for benign spinal tumors: theUniversity of California San Francisco preliminary experience. Technol Cancer Res Treat. 2007 Dec;6(6):595-604. doi: 10.1177/153303460700600602. PMID 17994789
- [Background] Dodd RL, Ryu MR, Kamnerdsupaphon P, Gibbs IC, Chang SD Jr, Adler JR Jr. CyberKnife radiosurgery for benign intradural extramedullary spinal tumors. Neurosurgery. 2006 Apr;58(4):674-85; discussion 674-85. doi: 10.1227/01.NEU.0000204128.84742.8F. PMID 16575331
- [Background] Schadev S, Dodd RL, Chang SD, Soltys SG, Adler JR, Luxton G, Choi CYH, Tupper LA, Gibbs IC. Stereotactic Radiosurgery Yields Long-term Control for Benign Intradural, Extramedullary Spine Tumors. Int J Radiat Oncol Biol Phys 2009; 75:101 (Abstract)
- [Background] Korones DN, Padowski J, Factor BA, Constine LS. Do children with optic pathway tumors have an increased frequency of other central nervous system tumors? Neuro Oncol. 2003 Apr;5(2):116-20. doi: 10.1093/neuonc/5.2.116. PMID 12672283